CLINICAL TRIAL: NCT05499130
Title: A 14 Week Phase 2b, Randomized, Double-Blind, Dose-Ranging Study to Determine the Pharmacokinetics, Efficacy, Safety and Tolerability of TEV-48574 in Adult Patients With Ulcerative Colitis or Crohn's Disease (RELIEVE UCCD)
Brief Title: A Study to Test the Effect of TEV-48574 in Moderate to Severe Ulcerative Colitis or Crohn's Disease
Acronym: RELIEVE UCCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48574-IMM-20036; 2021-006881-19 (EudraCT Number); 2024-511089-36-00 (Registry Identifier: Clinical Trials Information System)
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Crohn Disease; Colitis, Ulcerative
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- TEV-48574, 450 mg (UC) (Experimental): Administered by subcutaneous infusion for participants with UC
  Interventions: Drug: TEV-48574
- TEV-48574, 900 mg (UC) (Experimental): Administered by subcutaneous infusion for participants with UC
  Interventions: Drug: TEV-48574
- TEV-48574, 1800 mg (UC) (Experimental): Administered by subcutaneous infusion for participants with UC. This arm was discontinued with Amend 03.
  Interventions: Drug: TEV-48574
- TEV-48574, 450 mg (CD) (Experimental): Administered by subcutaneous infusion for participants with CD
  Interventions: Drug: TEV-48574
- TEV-48574, 900 mg (CD) (Experimental): Administered by subcutaneous infusion for participants with CD
  Interventions: Drug: TEV-48574
- TEV-48574, 1800 mg (CD) (Experimental): Administered by subcutaneous infusion for participants with CD. This arm was discontinued with Amend 03.
  Interventions: Drug: TEV-48574
- Placebo UC (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo
- Placebo CD (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-48574 — Subcutaneous infusion
  Other Names: duvakitug
  Arms: TEV-48574, 1800 mg (CD); TEV-48574, 1800 mg (UC); TEV-48574, 450 mg (CD); TEV-48574, 450 mg (UC); TEV-48574, 900 mg (CD); TEV-48574, 900 mg (UC)
Drug: Placebo — Matching Placebo
  Arms: Placebo CD; Placebo UC

SUMMARY:
The primary objective is to characterize the efficacy TEV-48574 in adult participants with IBD (moderate to severe Ulcerative Colitis (UC) or Crohn's Disease (CD)) as assessed by induction of clinical remission (UC) and endoscopic response (CD) at week 14.

Secondary objectives:

* To evaluate the efficacy of 2 different doses of TEV-48574 as assessed by multiple standard measures
* To evaluate the safety and tolerability of 2 different doses of TEV-48574
* To evaluate the immunogenicity of 2 different dioses of TEV-48574

The study will consist of a screening period of up to 6 weeks (42 days), a 14-week treatment period, and a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ulcerative Colitis (UC) or Crohn's Disease (CD) for ≥3 months
* The participant is able to communicate satisfactorily with the investigator and to participate in, and comply with, the requirements of the study
* The participant is able to understand the nature of the study and any potential hazards associated with participating in the study
* Women of non-childbearing potential who are either surgically (documented hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or congenitally sterile as assessed by a physician, or 1-year postmenopausal
* Male participants (including vasectomized) with women of childbearing potential (WOCBP) partners (whether pregnant or not) must use condoms after the first investigational medicinal product (IMP) administration and throughout the study or until 50 days after the last IMP dose, whichever is longer

NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has any concomitant conditions or treatments that could interfere with study conduct, influence the interpretation of study observations/results, or put the participant at increased risk during the study as judged by the investigator and/or the clinical study physician
* Diagnosis of indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, or microscopic coliti
* Participant has colonic dysplasia or neoplasia, toxic megacolon, primary sclerosing cholangitis, known non-passable colonic stricture, presence of colonic or small bowel stoma, presence of non-passable colonic or small bowel obstruction or resection preventing the endoscopy procedure, or fulminant colitis
* Presence of active enteric infections (positive stool culture) or a history of serious infection (requiring parenteral antibiotic and/or hospitalization) within 4 weeks prior to the first screening visit
* Participant anticipates requiring major surgery during this study.
* A participant is Hepatitis B core antibody or surface antigen positive and/or Hepatitis C antibody positive with detectable ribonucleic acids, or positive human immunodeficiency virus types 1 or 2 at screening.
* A history of an opportunistic infection (eg, cytomegalovirus retinitis, Pneumocystis carinii, or aspergillosis)
* A history of more than 2 herpes zoster episode in the last 5 years or multimetameric herpes zoster
* A history of or ongoing chronic or recurrent serious infectious disease (eg, infected indwelling prosthesis or osteomyelitis)
* The participant is currently pregnant or lactating or is planning to become pregnant or to lactate during the study or for at least 50 days after administration of the last dose of IMP in case of early termination. Any woman becoming pregnant during the study will be withdrawn from the study.
* Presence of a transplanted organ
* A history of malignancy within the last 5 years (exception: basal cell carcinoma or in situ carcinoma of the cervix if successful curative therapy occurred at least 12 months prior to screening) or curatively resected papillary thyroid cance
* Current or history (within 2 years) of serious psychiatric disease or alcohol or drug abuse
* Participants with incurable diseases, persons in nursing homes, and participants incapable of giving written informed consent

NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (164):
- United States (36):
  - Teva Investigational Site 15568, Sun City, Arizona
  - Teva Investigational Site 15556, San Diego, California
  - Teva Investigational Site 15747, San Diego, California
  - Teva Investigational Site 15357, Kissimmee, Florida
  - Teva Investigational Site 15563, Miami, Florida
  - Teva Investigational Site 15365, Miami, Florida
  - Teva Investigational Site 15748, Miami, Florida
  - Teva Investigational Site 15375, Orlando, Florida
  - Teva Investigational Site 15359, Pinellas Park, Florida
  - Teva Investigational Site 15566, Glenview, Illinois
  - Teva Investigational Site 15567, Gurnee, Illinois
  - Teva Investigational Site 15574, New Albany, Indiana
  - Teva Investigational Site 15362, Iowa City, Iowa
  - Teva Investigational Site 15367, Kansas City, Kansas
  - Teva Investigational Site 15368, Louisville, Kentucky
  - Teva Investigational Site 15575, Louisville, Kentucky
  - Teva Investigational Site 15363, Columbia, Maryland
  - Teva Investigational Site 15358, Liberty, Missouri
  - Teva Investigational Site 15373, St Louis, Missouri
  - Teva Investigational Site 15369, Las Vegas, Nevada
  - Teva Investigational Site 15558, North Massapequa, New York
  - Teva Investigational Site 15370, Chapel Hill, North Carolina
  - Teva Investigational Site 15750, Beavercreek, Ohio
  - Teva Investigational Site 15557, Greenville, South Carolina
  - Teva Investigational Site 15573, Cordova, Tennessee
  - Teva Investigational Site 15360, Austin, Texas
  - Teva Investigational Site 15371, Dallas, Texas
  - Teva Investigational Site 15569, Garland, Texas
  - Teva Investigational Site 15559, Harlingen, Texas
  - Teva Investigational Site 15366, Katy, Texas
  - Teva Investigational Site 15743, Lubbock, Texas
  - Teva Investigational Site 15372, Pearland, Texas
  - Teva Investigational Site 15374, San Antonio, Texas
  - Teva Investigational Site 15565, Southlake, Texas
  - Teva Investigational Site 15361, Tyler, Texas
  - Teva Investigational Site 15364, Salt Lake City, Utah
- Austria (2):
  - Teva Investigational Site 33055, Innsbruck
  - Teva Investigational Site 33056, Vienna
- Belgium (2):
  - Teva Investigational Site 37134, Edegem
  - Teva Investigational Site 37133, Liège
- Bulgaria (5):
  - Teva Investigational Site 59243, Gorna Oryahovitsa
  - Teva Investigational Site 59198, Pleven
  - Teva Investigational Site 59197, Sofia
  - Teva Investigational Site 59199, Sofia
  - Teva Investigational Site 59196, Sofia
- Teva Investigational Site 11257, Winnipeg, Manitoba, Canada
- Czechia (5):
  - Teva Investigational Site 54221, Brno
  - Teva Investigational Site 54222, Klatovy
  - Teva Investigational Site 54241, Prague
  - Teva Investigational Site 54220, Slaný
  - Teva Investigational Site 54242, Zábřeh
- France (4):
  - Teva Investigational Site 35280, Caen
  - Teva Investigational Site 35295, Nantes
  - Teva Investigational Site 35277, Nice
  - Teva Investigational Site 35279, Saint-Priest-en-Jarez
- Georgia (6):
  - Teva Investigational Site 81057, Tbilisi
  - Teva Investigational Site 81052, Tbilisi
  - Teva Investigational Site 81054, Tbilisi
  - Teva Investigational Site 81056, Tbilisi
  - Teva Investigational Site 81053, Tbilisi
  - Teva Investigational Site 81055, Tbilisi
- Germany (8):
  - Teva Investigational Site 32796, Berlin
  - Teva Investigational Site 32872, Berlin
  - Teva Investigational Site 32873, Duisburg
  - Teva Investigational Site 32793, Kiel
  - Teva Investigational Site 32797, Leipzig
  - Teva Investigational Site 32795, Tübingen
  - Teva Investigational Site 32794, Ulm
  - Teva Investigational Site 32874, Wipperfürth
- Hungary (5):
  - Teva Investigational Site 51334, Budapest
  - Teva Investigational Site 51335, Budapest
  - Teva Investigational Site 51336, Gyöngyös
  - Teva Investigational Site 51333, Székesfehérvár
  - Teva Investigational Site 51338, Vác
- Israel (5):
  - Teva Investigational Site 80179, Afula
  - Teva Investigational Site 80191, Beersheba
  - Teva Investigational Site 80184, Holon
  - Teva Investigational Site 80182, Kfar Saba
  - Teva Investigational Site 80180, Rehovot
- Italy (7):
  - Teva Investigational Site 30304, Brescia
  - Teva Investigational Site 30285, Milan
  - Teva Investigational Site 30286, Milan
  - Teva Investigational Site 30284, Rozzano
  - Teva Investigational Site 30303, San Donato Milanese
  - Teva Investigational Site 30300, San Giovanni Rotondo
  - Teva Investigational Site 30301, Turin
- Japan (9):
  - Teva Investigational Site 84112, Fukuoka
  - Teva Investigational Site 84110, Kashiwa
  - Teva Investigational Site 84118, Nagoya
  - Teva Investigational Site 84113, Osaka
  - Teva Investigational Site 84114, Sakura
  - Teva Investigational Site 84117, Tokyo
  - Teva Investigational Site 84116, Tokyo
  - Teva Investigational Site 84115, Tokyo
  - Teva Investigational Site 84111, Toyama
- Norway (2):
  - Teva Investigational Site 41015, Lorenskog
  - Teva Investigational Site 41014, Tromsø
- Poland (41):
  - Teva Investigational Site 53565, Bydgoszcz
  - Teva Investigational Site 53542, Częstochowa
  - Teva Investigational Site 53543, Elblag
  - Teva Investigational Site 53544, Gdansk
  - Teva Investigational Site 53545, Gdynia
  - Teva Investigational Site 53571, Jelenia Góra
  - Teva Investigational Site 53546, Katowice
  - Teva Investigational Site 53560, Krakow
  - Teva Investigational Site 53548, Krakow
  - Teva Investigational Site 53512, Krakow
  - Teva Investigational Site 53547, Kłodzko
  - Teva Investigational Site 53515, Lodz
  - Teva Investigational Site 53514, Lodz
  - Teva Investigational Site 53518, Nowy Targ
  - Teva Investigational Site 53559, Opole
  - Teva Investigational Site 53572, Piotrkow Trybunalski
  - Teva Investigational Site 53517, Poznan
  - Teva Investigational Site 53516, Poznan
  - Teva Investigational Site 53566, Poznan
  - Teva Investigational Site 53513, Rzeszów
  - Teva Investigational Site 53550, Sopot
  - Teva Investigational Site 53551, Staszów
  - Teva Investigational Site 53508, Szczecin
  - Teva Investigational Site 53519, Szczecin
  - Teva Investigational Site 53552, Tarnów
  - Teva Investigational Site 53573, Tarnów
  - Teva Investigational Site 53553, Torun
  - Teva Investigational Site 53554, Wadowice
  - Teva Investigational Site 53557, Warsaw
  - Teva Investigational Site 53570, Warsaw
  - Teva Investigational Site 53556, Warsaw
  - Teva Investigational Site 53555, Warsaw
  - Teva Investigational Site 53558, Wroclaw
  - Teva Investigational Site 53510, Wroclaw
  - Teva Investigational Site 53567, Wroclaw
  - Teva Investigational Site 53562, Wroclaw
  - Teva Investigational Site 53520, Wroclaw
  - Teva Investigational Site 53549, Wroclaw
  - Teva Investigational Site 53563, Wroclaw
  - Teva Investigational Site 53509, Zamość
  - Teva Investigational Site 53511, Łęczna
- Slovakia (8):
  - Teva Investigational Site 62098, Banská Bystrica
  - Teva Investigational Site 62074, Bardejov
  - Teva Investigational Site 62073, Bratislava
  - Teva Investigational Site 62071, Košice
  - Teva Investigational Site 62076, Prešov
  - Teva Investigational Site 62097, Prešov
  - Teva Investigational Site 62099, Rimavská Sobota
  - Teva Investigational Site 62072, Šahy
- Spain (7):
  - Teva Investigational Site 31325, Alicante
  - Teva Investigational Site 31302, Córdoba
  - Teva Investigational Site 31293, Huelva
  - Teva Investigational Site 31301, Las Palmas de Gran Canaria
  - Teva Investigational Site 31318, Santiago de Compostela
  - Teva Investigational Site 31291, Seville
  - Teva Investigational Site 31292, Valencia
- Ukraine (10):
  - Teva Investigational Site 58327, Chernivtsi
  - Teva Investigational Site 58324, Ivano-Frankivsk
  - Teva Investigational Site 58329, Lviv
  - Teva Investigational Site 58325, Lviv
  - Teva Investigational Site 58332, Lviv
  - Teva Investigational Site 58328, Ternopil
  - Teva Investigational Site 58322, Uzhhorod
  - Teva Investigational Site 58323, Uzhhorod
  - Teva Investigational Site 58330, Vinnytsia
  - Teva Investigational Site 58331, Vinnytsia
- Teva Investigational Site 34305, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please visit www.clinicalstudydatarequest.com to make your request

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this trial, 290 participants were randomized, and 286 participants were analyzed; 4 randomized participants (2 ulcerative colitis [UC] and 2 crohn's disease [CD]) were excluded from all analyses for non-compliance with Good Clinical Practice.
Pre-assignment Details: Participants were randomized to 1 of 4 treatment groups (TEV-48574 450 milligrams [mg], TEV-48574 900 mg, TEV-48574 1800 mg, or placebo to match TEV-48574) by indication UC and CD. The treatment arm TEV-48574 1800 mg was discontinued. Therefore, the participants randomized to TEV-48574 1800 mg arm were not included in the overall efficacy analysis for the trial (Modified Intent-to-treat [mITT] Analysis Set).
Groups:
- Placebo (UC): Participants with UC received placebo matched to TEV-48574 administered every 2 weeks (Q2W) (for a total of 7 doses) by subcutaneous (SC) injection during the 14-week treatment period.
- TEV-48574 450 mg (UC): Participants with UC received a single loading dose (2250 mg) of TEV-48574 by SC injection, followed by 6 induction doses (450 mg) of TEV-48574 Q2W by SC injection during the 14-week treatment period.
- TEV-48574 900 mg (UC): Participants with UC received a single loading dose (2250 mg) of TEV-48574 by SC injection, followed by 6 induction doses (900 mg) of TEV-48574 Q2W by SC injection during the 14-week treatment period.
- TEV-48574 1800 mg (UC): Participants with UC received a single loading dose (2250 mg) of TEV-48574 by SC injection, followed by 6 induction doses (1800 mg) of TEV-48574 Q2W by SC injection during the 14-week treatment period.
- Placebo (CD): Participants with CD received placebo matched to TEV-48574 administered Q2W (for a total of 7 doses) by SC injection during the 14-week treatment period.
- TEV-48574 450 mg (CD): Participants with CD received a single loading dose (2250 mg) of TEV-48574 by SC injection, followed by 6 induction doses (450 mg) of TEV-48574 Q2W by SC injection during the 14-week treatment period.
- TEV-48574 900 mg (CD): Participants with CD received a single loading dose (2250 mg) of TEV-48574 by SC injection, followed by 6 induction doses (900 mg) of TEV-48574 Q2W by SC injection during the 14-week treatment period.
- TEV-48574 1800 mg (CD): Participants with CD received a single loading dose (2250 mg) of TEV-48574 by SC injection, followed by 6 induction doses (1800 mg) of TEV-48574 Q2W by SC injection during the 14-week treatment period.
Period: Overall Study
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC) | TEV-48574 1800 mg (UC) | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD) | TEV-48574 1800 mg (CD)
Started | 44 | 47 | 46 | 7 | 46 | 46 | 47 | 3
Received at Least 1 Dose of Study Drug | 44 | 47 | 46 | 7 | 46 | 46 | 46 | 3
mITT Analysis Set (The mITT analysis set for each indication (UC or CD) included only those participants who received at least 1 dose of placebo, TEV-48574 low dose, or TEV-48574 medium dose.) | 44 | 47 | 46 | 0 | 46 | 46 | 46 | 0
Immunogenicity Analysis Set (The immunogenicity analysis set included all participants in all randomized participants who received at least 1 dose of TEV-48574 and who had at least 1 reportable immunogenicity result.) | 0 | 47 | 45 | 7 | 0 | 46 | 46 | 3
Completed | 39 | 47 | 45 | 7 | 37 | 37 | 43 | 3
Not Completed | 5 | 0 | 1 | 0 | 9 | 9 | 4 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 1 | 4 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 5 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Other Than Specified | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set for each indication (UC or CD) included all randomized participants.
Groups:
- Placebo (UC): Participants with UC received placebo matched to TEV-48574 administered Q2W (for a total of 7 doses) by SC injection during the 14-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC) | TEV-48574 1800 mg (UC) | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD) | TEV-48574 1800 mg (CD) | Total
Number analyzed (Participants) | 44 | 47 | 46 | 7 | 46 | 46 | 47 | 3 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (13.08) | 38.7 (12.99) | 42.1 (13.19) | 40.9 (16.24) | 38.3 (15.13) | 42.5 (15.08) | 38.1 (13.58) | 43.7 (23.54) | 40.4 (13.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 19 | 5 | 24 | 19 | 16 | 1 | 116
  Male | 30 | 29 | 27 | 2 | 22 | 27 | 31 | 2 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 6
  Not Hispanic or Latino | 42 | 46 | 45 | 7 | 46 | 43 | 46 | 3 | 278
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 6
  Race: Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 4
  Race: White | 43 | 44 | 45 | 7 | 45 | 45 | 41 | 3 | 273
  Race: Other | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Race: Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Modified Mayo Score (MMS) [Mean (Standard Deviation); unit: units on a scale] — The MMS is a tool designed to measure disease activity for UC. It consisted of 3 subscores: stool frequency, rectal bleeding and endoscopic subscore as determined during central review. Each subscore was graded from 0 (normal) to 3 (severe). These individual subscores were summed up to give a total MMS ranging from 0 (normal or inactive disease) to 9 (severe disease), where higher scores indicated more severe disease activity. Population: Number analyzed = participants with UC.
  units on a scale
    number analyzed (Participants) | 44 | 47 | 46 | 7 | 0 | 0 | 0 | 0 | 144
    (all) | 6.8 (1.16) | 6.6 (1.15) | 6.8 (1.11) | 6.6 (1.13) |  |  |  |  | 6.7 (1.14)
Simple Endoscopic Score for Crohn's Disease (SES-CD) [Mean (Standard Deviation); unit: units on a scale] — SES-CD assesses following 4 components: presence of ulcers and strictures, percentage of ulcerated surfaces and affected surface. Each of these components scored on a scale of 0 (none/unaffected) to 3 (worst). Each of these 4 components was assessed in 5 segments: rectum, sigmoid and left colon, transverse colon, right colon, and ileum. SES-CD was the sum of individual scores of each components across 5 segments. Range of SES-CD scores was 0 (none) - 12 (severe) for each segment, and 0 (none) - 60 (severe) for overall SES-CD score, with larger scores indicating greater degree of inflammation. Population: Number analyzed = participants with CD.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 46 | 46 | 47 | 3 | 142
    (all) |  |  |  |  | 12.0 (5.70) | 12.7 (6.64) | 12.1 (5.81) | 7.7 (2.89) | 12.1 (6.01)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Moderate to Severe UC Who Showed Clinical Remission as Defined by the MMS
Description: The MMS is a tool designed to measure disease activity for UC. It consisted of 3 subscores: stool frequency, rectal bleeding and endoscopic subscore as determined during central review. Each subscore was graded from 0 (normal) to 3 (severe). These individual subscores were summed up to give a total MMS ranging from 0 (normal or inactive disease) to 9 (severe disease), where higher scores indicated more severe disease activity. Clinical remission was defined as MMS ≤2 points with Mayo stool frequency subscore of 0 or 1, Mayo rectal bleeding subscore of 0, and centrally read endoscopic score of 0 or 1, where a score of 1 did not include "friability".
Time Frame: Week 14
Population: The mITT analysis set for UC included only those participants who received at least 1 dose of placebo, TEV-48574 450 mg, or TEV-48574 900 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC)
Number analyzed (Participants) | 44 | 47 | 46
Participants | 9 | 17 | 22
Statistical Analysis 1: Comparison: Placebo (UC) vs TEV-48574 450 mg (UC); Test type: Other; Difference in Response Rate = 15.7
Statistical Analysis 2: Comparison: Placebo (UC) vs TEV-48574 450 mg (UC); Test type: Other; Posterior Probability = 0.949 — A beta-binomial model was employed to obtain this posterior probability using a non-informative prior to assess superior efficacy compared to placebo
Statistical Analysis 3: Comparison: Placebo (UC) vs TEV-48574 900 mg (UC); Test type: Other; Difference in Response Rate = 27.4
Statistical Analysis 4: Comparison: Placebo (UC) vs TEV-48574 900 mg (UC); Test type: Other; Posterior Probability = 0.997 — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Number of Participants With Moderate to Severe CD Who Showed an Endoscopic Response as Defined by the SES-CD
Description: The SES-CD assessed the degree of inflammation. The SES-CD assesses the following 4 components: presence of ulcers, percentage of ulcerated surfaces, affected surface, and presence of strictures. Each of these components was scored on a scale of 0 (none/unaffected) to 3 (worst). In the SES-CD, each of these 4 components was assessed in the 5 segments: the rectum, sigmoid and left colon, transverse colon, right colon, and ileum. The SES-CD was the sum of the individual scores of each of the components across the 5 segments. The range of SES-CD scores was 0 (none) - 12 (severe) for each segment, and 0 (none) - 60 (severe) for the overall SES-CD score, with larger scores indicating greater degree of inflammation. Endoscopic response at Week 14 in participants with moderate to severe CD was defined as a reduction in SES-CD of at least 50% from baseline.
Time Frame: Baseline to Week 14
Population: The mITT analysis set for CD included only those participants who received at least 1 dose of placebo, TEV-48574 450 mg, or TEV-48574 900 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD)
Number analyzed (Participants) | 46 | 46 | 46
Participants | 6 | 12 | 22
Statistical Analysis 1: Comparison: Placebo (CD) vs TEV-48574 450 mg (CD); Test type: Other; Difference in Response Rate = 13.0
Statistical Analysis 2: Comparison: Placebo (CD) vs TEV-48574 450 mg (CD); Test type: Other; Posterior Probability = 0.939 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo (CD) vs TEV-48574 900 mg (CD); Test type: Other; Difference in Response Rate = 34.8
Statistical Analysis 4: Comparison: Placebo (CD) vs TEV-48574 900 mg (CD); Test type: Other; Posterior Probability = 1.000 — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Number of Participants With Moderate to Severe UC With a Clinical Response as Defined by the MMS
Description: The MMS is a tool designed to measure disease activity for UC. It consisted of 3 subscores: stool frequency, rectal bleeding and endoscopic subscore as determined during central review. Each subscore was graded from 0 (normal) to 3 (severe). These individual subscores were summed up to give a total MMS ranged from 0 (normal or inactive disease) to 9 (severe disease), where higher scores indicated more severe disease activity. Clinical response was defined as a decrease from baseline in the MMS of at least 2 points and at least a 30% reduction from baseline with either a decrease in rectal bleeding subscore of at least 1 or an absolute rectal bleeding subscore of ≤1.
Time Frame: Baseline to Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC)
Number analyzed (Participants) | 44 | 47 | 46
Participants | 23 | 38 | 32

4. Secondary Outcome: Number of Participants With Moderate to Severe UC With Endoscopic Improvement as Defined by the Mayo Endoscopic Subscore (MES)
Description: The endoscopic subscore evaluation for the MMS consisted of independent, blinded, central review of a high-resolution recorded video. The endoscopic subscore assessed disease activity from 0 (normal or inactive disease) to 3 (severe activity). Higher scores indicated more severe disease activity. Endoscopic improvement was defined as a MES of 0 or 1 at Week 14.
Time Frame: Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC)
Number analyzed (Participants) | 44 | 47 | 46
Participants | 10 | 21 | 23

5. Secondary Outcome: Number of Participants With Moderate to Severe UC With Endoscopic Remission as Defined by the MES
Description: The endoscopic subscore evaluation for the MMS consisted of independent, blinded, central review of a high-resolution recorded video. The endoscopic subscore assessed disease activity from 0 (normal or inactive disease) to 3 (severe activity). Higher scores indicated more severe disease activity. Endoscopic remission was defined as a MES of 0 at Week 14.
Time Frame: Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC)
Number analyzed (Participants) | 44 | 47 | 46
Participants | 3 | 8 | 8

6. Secondary Outcome: Number of Participants With Moderate to Severe UC With a Clinical Response as Defined by 2-item Patient-reported Outcome (PRO2) Score
Description: The PRO2-UC score was derived from 2 parameters from the MMS: stool frequency and rectal bleeding, recorded daily by the participant using a handheld electronic diary over each of the preceding 7 days. Each parameter ranged from 0 (normal) to 3 (severe) with each subscore representing an average over the preceding 7 days. The total score was the summation of the subscores and therefore ranged from 0 (normal or inactive disease) to 6 (severe activity), where higher scores indicated more severe disease activity. Clinical response was defined as decrease from baseline of at least 50% in PRO2 (stool frequency and rectal bleeding) at Week 14.
Time Frame: Baseline to Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC)
Number analyzed (Participants) | 44 | 47 | 46
Participants | 22 | 39 | 34

7. Secondary Outcome: Number of Participants With Moderate to Severe UC With a Clinical Remission as Defined by PRO2 Score
Description: The PRO2-UC score was derived from 2 parameters from the MMS: stool frequency and rectal bleeding, recorded daily by the participant using a handheld electronic diary over each of the preceding 7 days. Each parameter ranged from 0 (normal) to 3 (severe) with each subscore representing an average over the preceding 7 days. The total score was the summation of the subscores and therefore ranged from 0 (normal or inactive disease) to 6 (severe activity), where higher scores indicated more severe disease activity. Clinical remission was defined as score of stool frequency = 0 and rectal bleeding = 0 on the PRO2 scale at Week 14.
Time Frame: Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC)
Number analyzed (Participants) | 44 | 47 | 46
Participants | 4 | 14 | 11

8. Secondary Outcome: Number of Participants With Moderate to Severe CD With an Endoscopic Response as Defined by the Modified Multiplier-Simple Endoscopic Score (MM-SES-CD)
Description: The MM-SES-CD is an endoscopic scoring tool that considers each individual parameter's prognostic value for achieving endoscopic remission while on active therapy. The SES-CD assesses the following 4 components: presence of ulcers, percentage of ulcerated surfaces, affected surface, and presence of strictures. Each of these components was scored on a scale of 0 (none/unaffected) to 3 (worst). In the SES-CD, each of these 4 components was assessed in the 5 segments: the rectum, sigmoid and left colon, transverse colon, right colon, and ileum. The SES-CD was the sum of the individual scores of each of the components across the 5 segments. The range of SES-CD scores was 0 (none) - 12 (severe) for each segment, and 0 (none) - 60 (severe) for the overall SES-CD score, with higher scores indicating a greater degree of inflammation. Endoscopic response was defined as a decrease in MM-SES-CD of ≥50% from baseline at Week 14.
Time Frame: Baseline to Week 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD)
Number analyzed (Participants) | 46 | 46 | 46
Participants | 6 | 16 | 18

9. Secondary Outcome: Number of Participants With Moderate to Severe CD With a Clinical Response as Defined by Crohn's Disease Activity Index (CDAI) Score
Description: The CDAI score consisted of an adjusted composite sum of 8 parameters, including daily diary evaluation for severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight, and hematocrit. The subscores of abdominal pain (0 [no pain] to 3 [worst pain]), general well-being (0 [well] to 4 [terrible]), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score that ranged from 0 (none) to 600 (severe) with a higher score indicating a worse outcome. Clinical response was defined as a ≥100-point decrease in CDAI score from baseline.
Time Frame: Baseline to Weeks 4, 8, 12 and 14
Population: The mITT analysis set for CD included only those participants who received at least 1 dose of placebo, TEV-48574 450 mg, or TEV-48574 900 mg. Here, 'number analyzed' = participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD)
Number analyzed (Participants) | 46 | 46 | 46
Participants
  Week 4: number analyzed (Participants) | 40 | 45 | 44
  Week 4 | 15 | 24 | 18
  Week 8: number analyzed (Participants) | 44 | 46 | 46
  Week 8 | 19 | 30 | 25
  Week 12: number analyzed (Participants) | 45 | 46 | 45
  Week 12 | 22 | 31 | 31
  Week 14 | 24 | 30 | 30

10. Secondary Outcome: Number of Participants With Moderate to Severe CD With a Clinical Remission as Defined by CDAI Score
Description: The CDAI score consisted of an adjusted composite sum of 8 parameters, including daily diary evaluation for severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight, and hematocrit. The subscores of abdominal pain (0 [no pain] to 3 [worst pain]), general well-being (0 [well] to 4 [terrible]), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score that ranged from 0 (none) to 600 (severe) with a higher score indicating a worse outcome. Clinical remission was defined as a CDAI score <150 at Week 14.
Time Frame: Week 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD)
Number analyzed (Participants) | 46 | 46 | 46
Participants | 19 | 23 | 25

11. Secondary Outcome: Number of Participants With Moderate to Severe CD With a Clinical Response as Defined by PRO2-CD Score
Description: The PRO2-CD score was the sum of the daily stool frequency subscore (0 [normal] to 3 [severe]) and abdominal pain subscore (0 [no pain] to 3 [worst pain]) from the CDAI. Total PRO2-CD score ranged from 0 (normal) - 6 (severe), with higher scores indicating more severe disease. These were recorded daily by the participant using a handheld electronic diary over each of the preceding 7 days. Clinical response was defined as a decrease from baseline of at least 50% in PRO2-CD (abdominal pain and stool frequency) at Week 14.
Time Frame: Baseline to Week 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD)
Number analyzed (Participants) | 46 | 46 | 46
Participants | 8 | 16 | 14

12. Secondary Outcome: Number of Participants With Moderate to Severe CD With a Clinical Remission as Defined by PRO2-CD Score
Description: The PRO2-CD score was the sum of the daily stool frequency subscore (0 [normal] to 3 [severe]) and abdominal pain subscore (0 [no pain] to 3 [worst pain]) from the CDAI. Total PRO2-CD score ranged from 0 (normal) - 6 (severe), with higher scores indicating more severe disease. These were recorded daily by the participant using a handheld electronic diary over each of the preceding 7 days. Clinical remission was defined as abdominal pain ≤1 and stool frequency ≤3 on the PRO2-CD scale at Week 14
Time Frame: Week 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD)
Number analyzed (Participants) | 46 | 46 | 46
Participants | 12 | 17 | 17

13. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs were considered TEAEs if onset occurred on or after the first dose date. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 1) up to Week 18
Population: The safety analysis set for each indication (UC or CD) included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC) | TEV-48574 1800 mg (UC) | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD) | TEV-48574 1800 mg (CD)
Number analyzed (Participants) | 44 | 47 | 46 | 7 | 46 | 46 | 46 | 3
Participants | 23 | 23 | 20 | 2 | 22 | 31 | 20 | 2

14. Secondary Outcome: Number of Participants Who Stopped Taking the Investigational Medicinal Product (IMP) Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 1) up to Week 18
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC) | TEV-48574 1800 mg (UC) | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD) | TEV-48574 1800 mg (CD)
Number analyzed (Participants) | 44 | 47 | 46 | 7 | 46 | 46 | 46 | 3
Participants | 2 | 0 | 1 | 0 | 1 | 4 | 1 | 0

15. Secondary Outcome: Number of Participants With Treatment-emergent Anti-Drug Antibodies (ADAs)
Description: Treatment-emergent ADA positive: - the participant had a positive ADA sample (after first dose of study drug) but not at baseline (prior to first dose of study drug), or - the participant had a positive ADA sample at baseline (prior to first dose of study drug) and at the visit (after first dose of study drug), with at least a 4-fold increase in titer level.
Time Frame: Weeks 2, 4, 8, 14, and 18
Population: The immunogenicity analysis set included all randomized participants who received at least 1 dose of TEV-48574 and who had at least 1 reportable immunogenicity result.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC) | TEV-48574 1800 mg (UC) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD) | TEV-48574 1800 mg (CD)
Number analyzed (Participants) | 47 | 45 | 7 | 46 | 46 | 3
Participants
  Week 2 | 0 | 0 | 0 | 4 | 1 | 0
  Week 4 | 0 | 2 | 0 | 2 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14 | 0 | 0 | 0 | 0 | 0 | 0
  Week 18 | 1 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of ADA Positive Participants With the Presence of Neutralizing ADA
Description: as for outcome 15
Time Frame: Weeks 2, 4, 8, 14, and 18
Population: The immunogenicity analysis set included all randomized participants who received at least 1 dose of TEV-48574 and who had at least 1 reportable immunogenicity result. 'Overall number of participants analyzed' = ADA positive participants. 'Number analyzed' = ADA positive participants at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC) | TEV-48574 1800 mg (UC) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD) | TEV-48574 1800 mg (CD)
Number analyzed (Participants) | 1 | 2 | 0 | 4 | 1 | 0
Participants
  Week 2: number analyzed (Participants) | 0 | 0 | 0 | 4 | 1 | 0
  Week 2 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 0 | 2 | 0 | 2 | 0 | 0
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Week 14 | 0 | 0 | 0 | 0 | 0 | 0
  Week 18: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Week 18 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Week 18
Description: The safety analysis set for each indication (UC or CD) included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo (UC) | TEV-48574 450 mg (UC) | TEV-48574 900 mg (UC) | TEV-48574 1800 mg (UC) | Placebo (CD) | TEV-48574 450 mg (CD) | TEV-48574 900 mg (CD) | TEV-48574 1800 mg (CD)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/47 | 0/46 | 0/7 | 0/46 | 0/46 | 0/46 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/47 | 1/46 | 0/7 | 5/46 | 6/46 | 1/46 | 0/3
Other Adverse Events (participants affected / at risk) | 6/44 | 10/47 | 6/46 | 2/7 | 9/46 | 9/46 | 5/46 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (UC) (N=44) | TEV-48574 450 mg (UC) (N=47) | TEV-48574 900 mg (UC) (N=46) | TEV-48574 1800 mg (UC) (N=7) | Placebo (CD) (N=46) | TEV-48574 450 mg (CD) (N=46) | TEV-48574 900 mg (CD) (N=46) | TEV-48574 1800 mg (CD) (N=3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure orthostatic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Noninfective oophoritis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (UC) (N=44) | TEV-48574 450 mg (UC) (N=47) | TEV-48574 900 mg (UC) (N=46) | TEV-48574 1800 mg (UC) (N=7) | Placebo (CD) (N=46) | TEV-48574 450 mg (CD) (N=46) | TEV-48574 900 mg (CD) (N=46) | TEV-48574 1800 mg (CD) (N=3)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The treatment arm TEV-48574 1800 mg was discontinued. Therefore, the participants randomized to TEV-48574 1800 mg arm were not included in the overall efficacy analysis for the trial (mITT Analysis Set).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT05499130/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT05499130/SAP_001.pdf